CLINICAL TRIAL: NCT00091689
Title: Safety and Efficacy of an Immune Response Modifier to Treat Inoperable Advanced Melanoma Skin Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1501-852A
Record Dates: First submitted 2004-09-15; First posted 2004-09-17 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Melanoma
Keywords: Advanced Metastatic Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Drug: 852A

SUMMARY:
Study 1501-852A is a Phase 1 Study with the objective of determining safety and the highest tolerated dose of an immune response modifier cream directly applied to advanced, inoperable, melanoma skin lesions. The study will also measure blood levels of the drug and examine the potential anti-tumor activity of the cream.

ELIGIBILITY:
Inclusion Criteria:

* Have melanoma cutaneous metastasis or lentigo maligna melanoma unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Have a life expectancy of 4 months
* Have normal organ and bone marrow function

Exclusion Criteria:

* Need for non-steroidal anti-inflammatory drugs (NSAIDs) during the study
* Have a body mass index (BMI)> 30 kg/m2
* Have a history of, or clinical evidence of, myocardial ischemia, congestive heart failure, or myocardial arrhythmias requiring treatment within the past 6 months
* Have uncontrolled intercurrent or chronic illness, but not limited to, ongoing or active infection such as hepatitis B or C, immune dysfunction such as autoimmune disease, endocrine dysfunction such as hypo- or hyperthyroidism, psychiatric illness such as depression or suicidal tendency or social situations that would limit compliance with study requirements
* Have a history of disease requiring ongoing steroid treatment
* Have a history of seizure disorder (other than febrile seizures in childhood)
* Have a history of clinically significant coagulation or bleeding disorders or abnormalities
* Are HIV positive. HIV positive subjects are excluded from the study because of possible interactions with the immunomodulatory effects of 852A and because of potential pharmacokinetic interactions associated with combination retroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma